CLINICAL TRIAL: NCT01799018
Title: Role of Proteomics and Metallomics in Cerebral Vasospasm Following Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#225490
Record Dates: First submitted 2012-12-12; First posted 2013-02-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm; Hydrocephalus
Keywords: Xanthine Oxidase; Cerebrospinal fluid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid (CSF)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SAH Patients: Patients admitted with the diagnosis of aneurismal subarachnoid hemorrhage (SAH) and cerebral angiogram negative SAH who would need to have the external ventricular drain (EVD) placed for the management of hydrocephalus.
- Control Patients: Patients with non-hemorrhagic brain pathology such as posterior fossa tumor or stroke who will have the CSF sampling for diagnostic or therapeutic purposes.

SUMMARY:
The purpose of this study is to determine the role of Proteomics and Metallomics in Cerebral Vasospasm following Subarachnoid Hemorrhage

ELIGIBILITY:
Inclusion Criteria:

* Non traumatic SAH documented by CT scan
* Patient with SAH who would need external ventricular drain (EVD) for the management of hydrocephalus
* Patients with normal pressure Hydrocephalus that require an external drain
* Control (non - hemorrhagic) group - CSF collected from patients with posterior fossa tumor or stroke with EVD in place for the management of hydrocephalus.

Exclusion Criteria:

* Recent infection within last 1 month of presentation- can increase inflammatory markers
* Recent surgery or acute myocardial infarction within last 1 month of presentation
* Age > 89 years or < 18 years

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to University Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Protein identification and concentration | For the duration of CSF drainage, or until the 21st day after admission.
Metal ion identification and concentration | For the duration of CSF drainage, or until the 21st day after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Deshaies, MD, Principal Investigator — SUNY Upstate Medical University - Neurosurgery
Locations (1):
- State University of New York Upstate Medical University, Syracuse, New York, United States